CLINICAL TRIAL: NCT00004400
Title: Phase II Randomized Study of Physiologic Testosterone Replacement in Premenopausal, HIV-Positive Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13251; CDUMS-FDR001397
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-05

CONDITIONS: HIV Infections; Cachexia
Keywords: cachexia; disease-related problem/condition; human immunodeficiency virus infection; immunologic disorders and infectious disorders; nutrition; quality of life; rare disease; viral infection
MeSH Terms: conditions — HIV Infections; Cachexia; Acquired Immunodeficiency Syndrome; Immune System Diseases; Communicable Diseases; Rare Diseases; Virus Diseases | interventions — Testosterone

INTERVENTIONS:
Drug: testosterone

SUMMARY:
OBJECTIVES: I. Determine whether physiologic testosterone replacement can increase fat-free mass, therefore contributing to weight maintenance, improved muscle function, and quality of life in HIV-infected women.

II. Examine the mechanism of testosterone-induced increase in fat-free mass.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled study. Patients are randomized to one of three arms.

Arm I: Patients receive two placebo transdermal patches applied twice a week (every 3-4 days).

Arm II: Patients receive one testosterone transdermal patch and one placebo transdermal patch applied twice a week (every 3-4 days).

Arm III: Patients receive two testosterone transdermal patches applied twice a week (every 3-4 days).

Patients receive 12 weeks of treatment in the absence of adverse reaction or health deterioration. Patients are followed on day 1, every 2 weeks during treatment, and at the end of the recovery period. Quality of life is assessed before treatment begins and at weeks 6 and 12.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Histologically confirmed premenopausal HIV-positive women who have experienced 5-15% weight loss

--Prior/Concurrent Therapy--

* Endocrine therapy: At least 3 months since megestrol At least 3 months since anabolic or androgenic steroids At least 3 months since oral contraceptives At least 3 months since Depo-Provera No concurrent hormone replacement therapy
* Other: Concurrent retroviral or protease inhibitors allowed, dosage must be stable At least 3 months since ketoconazole At least 6 weeks since the initiation of protease inhibitors

--Patient Characteristics--

* Hepatic: No significant liver disease SGOT/SGPT no greater than 3 times upper limit of normal (ULN) Alkaline phosphatase no greater than 3 times ULN Bilirubin no greater than 2 mg/dL No medical complications due to alcohol abuse
* Renal: Not specified
* Cardiovascular: No significant cardiovascular disease No uncontrolled hypertension
* Other: Testosterone level (early morning) less than 30 ng/dL Normal gastrointestinal function as indicated by: Absence of diarrhea Normal D-xylose absorption test No acute opportunistic infections or infectious illness No malignant disease No history of breast cancer No history of endometrial cancer No fever of known or unknown origin No unremitting diarrhea defined as: At least 4 watery stools per day OR More than 4 watery stools recently OR Acute change in stool habit with fever No significant respiratory disease No diabetes No illicit drugs within the past 6 months No history of hyperandrogenic disorders such as: Hirsutism Polycystic ovary disease Not pregnant or lactating

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 1997-04; Study Completion 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, Study Chair — Charles Drew University of Medicine and Science
Locations (3):
- United States (3):
  - Charles R. Drew University of Medicine and Science, Los Angeles, California
  - Los Angeles County Harbor-UCLA Medical Center, Torrance, California
  - Washington University School of Medicine, St Louis, Missouri